CLINICAL TRIAL: NCT04453696
Title: Dentist-Patient Communication on Dental Anxiety Using the Social Media and Timing in Communication: A Double-blinded Randomized Controlled Trial
Brief Title: Dentist-Patient Communication on Dental Anxiety Using the Social Media and Timing in Communication
Status: Completed | Type: Observational
Sponsor: Karadeniz Technical University (Other)
Collaborators: Onur Yilmaz (Unknown); Pinar Sivrikaya (Unknown)
Responsible Party: Principal Investigator, Efe Sivrikaya, Assistant Prof., Karadeniz Technical University
Other Study IDs: KaradenizTU01
Record Dates: First submitted 2020-06-11; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Dental Anxiety; Timing in Dentist-Patient Communication
Keywords: Communication; Dental anxiety; Social Media
MeSH Terms: conditions — Communication

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Communication before operation: Communication was established before the operation.
  Interventions: Behavioral: Assessment scales-the Spielberger's State-Trait Anxiety Inventory, Modified Dental Anxiety Scale and a visual analog scale.
- Communication after operation: Communication was established after the operation.
  Interventions: Behavioral: Assessment scales-the Spielberger's State-Trait Anxiety Inventory, Modified Dental Anxiety Scale and a visual analog scale.
- Communication before and after operation: Communication took place both before and after the operation.
  Interventions: Behavioral: Assessment scales-the Spielberger's State-Trait Anxiety Inventory, Modified Dental Anxiety Scale and a visual analog scale.
- No communication: No communication.
  Interventions: Behavioral: Assessment scales-the Spielberger's State-Trait Anxiety Inventory, Modified Dental Anxiety Scale and a visual analog scale.

INTERVENTIONS:
Behavioral: Assessment scales-the Spielberger's State-Trait Anxiety Inventory, Modified Dental Anxiety Scale and a visual analog scale. — STAI-S, like kinetic energy, refers to a palpable reaction or process taking place at a given time and level of intensity. STAI-T, like potential energy, refers to individual differences in reactions. Both of STAI-S and STAI-T scales includes 20 questions. For each question, the scores range from 1 (almost never) to 4 (almost always) points. For both scales, the sum of the scores ranges from 20 to 80. A score between 36 and 41 refers to a mean anxiety level, with values greater than 41 classified as a high level of anxiety.
  The MDAS consists of 5 questions that measure anxiety at different stages of dental treatment. The options range from 1 (not anxious) to 5 (very anxious) for each question. The sum of the scores varies from 5 to 25; values between 19 and 25 indicate a high level of dental anxiety.
  The VAS scale was included in the present study to determine how anxious the patients felt according to their own thoughts. Scores range from 0 (no anxiety) to 10 (extreme anxiety).

SUMMARY:
Scales application one week before and one week after impacted tooth extraction.

DETAILED DESCRIPTION:
The purpose of the present study was to assess the effects of dentist-patient communication via social media on dental anxiety, and second, to evaluate the appropriate timing of such communications.

Instagram's quick replies system was used to answer patients' questions to alleviate dental anxiety for patients undergoing impacted mandibular third-molar extraction under local anesthesia. Patients were assigned randomly into four groups according to timing of such communications: Communication before operation (n=36), Communication after operation (n=35), Communication before and after operation (n=36), and a control group who received no communication on social media (n=36). Dental anxiety was evaluated one week before and after the surgical operation using recognized assessment scales-the Spielberger's State-Trait Anxiety Inventory, Modified Dental Anxiety Scale and a visual analog scale.

ELIGIBILITY:
Inclusion Criteria:

* Must be able to use the Instagram platform. I
* Clinicial diagnosis of mesioangular impacted lower third molar according to the classification of Winter and the Pell and Gregory classification (2 or 3/B).

Exclusion Criteria:

* Patients who previously obtained information from social media
* Bad dental history
* Systemic disease
* Pregnant

Ages: 22 Years to 36 Years | Sex: All
Age Groups: Adult
Study Population: The patients scheduled to undergo impacted lower third molar removal at the oral and maxillofacial surgery clinic at Karadeniz Teknik University were selected by randomly between 2018 and 2020
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2020-03-08 (Actual); Study Completion 2020-05-10 (Actual)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | 2 weeks
  The VAS scale was included in the present study to determine how anxious the patients felt according to their own thoughts. Scores range from 0 (no anxiety) to 10 (extreme anxiety).

OTHER OUTCOMES:
State-Trait Anxiety Inventory (STAI-T and STAI-S) | 2 weeks
  STAI-S, like kinetic energy, refers to a palpable reaction or process taking place at a given time and level of intensity. STAI-T, like potential energy, refers to individual differences in reactions. Both of STAI-S and STAI-T scales includes 20 questions. For each question, the scores range from 1 (almost never) to 4 (almost always) points. For both scales, the sum of the scores ranges from 20 to 80. A score between 36 and 41 refers to a mean anxiety level, with values greater than 41 classified as a high level of anxiety.
Modified Dental Anxiety Scale (MDAS) | 2 weeks
  The MDAS consists of 5 questions that measure anxiety at different stages of dental treatment. The options range from 1 (not anxious) to 5 (very anxious) for each question. The sum of the scores varies from 5 to 25; values between 19 and 25 indicate a high level of dental anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Efe Can Sivrikaya, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT04453696/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/96/NCT04453696/ICF_001.pdf